CLINICAL TRIAL: NCT06404203
Title: Investigation of the Effect of Oral Use of Lyophilised Royal Jelly (Apis Mellifera) on Cognitive Functions and Inflammation-Related Immune System Cytokine Levels in Elderly Individuals: A Randomized Controlled Trial
Brief Title: The Effect of Oral Use of Lyophilised Royal Jelly on Cognitive Functions and Immune System in Elderly Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Muhammet Ali Behesti BAYLAN, Assistant of Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: E-95961207-604.01.01-5745
Record Dates: First submitted 2023-07-09; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-07

CONDITIONS: Cognitive Change
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Royal Jelly 500 mg (Experimental): 30 volunteer
  Interventions: Dietary Supplement: Balparmak Apitera Royal Jelly Herbal Capsule Food Supplement 500 mg/day
- Royal Jelly 1000 mg (Experimental): 30 volunteer
  Interventions: Dietary Supplement: Balparmak Apitera Royal Jelly Herbal Capsule Food Supplement 1000 mg/day
- Royal Jelly 1500 mg (Experimental): 30 volunteer
  Interventions: Dietary Supplement: Balparmak Apitera Royal Jelly Herbal Capsule Food Supplement 1500 mg/day
- Placebo (Placebo Comparator): 30 volunteer
  Interventions: Other: Plasebo

INTERVENTIONS:
Dietary Supplement: Balparmak Apitera Royal Jelly Herbal Capsule Food Supplement 500 mg/day — Volunteers will receive Balparmak Apitera Royal Jelly Herbal Capsule Food Supplement in a dose of 500 mg/day for 4 weeks.
  Arms: Royal Jelly 500 mg
Dietary Supplement: Balparmak Apitera Royal Jelly Herbal Capsule Food Supplement 1000 mg/day — Volunteers will receive Balparmak Apitera Royal Jelly Herbal Capsule Food Supplement in a dose of 10000 mg/day for 4 weeks.
  Arms: Royal Jelly 1000 mg
Dietary Supplement: Balparmak Apitera Royal Jelly Herbal Capsule Food Supplement 1500 mg/day — Volunteers will receive Balparmak Apitera Royal Jelly Herbal Capsule Food Supplement in a dose of 1500 mg/day for 4 weeks.
  Arms: Royal Jelly 1500 mg
Other: Plasebo — Volunteers will receive a soft vegan gelatin capsule containing lactose in a dose of 1500 mg/day for 4 weeks.
  Arms: Placebo

SUMMARY:
Dementia is a significant public health problem, affecting 47 million people worldwide in 2015, according to World Health Organization data. It is expected to increase to 75 million in 2030 and reach 132 million in 2050.

Royal jelly is used as a supplement in treating of cancer, hypertension, diabetes and neurodegenerative diseases due to its antioxidant, anti-inflammatory, neuroprotective, cardioprotective, anti-proliferative and anti-fatigue properties. There are preclinical studies on the curative and protective effects of royal jelly on cognitive functions.

This randomized controlled, double-blind clinical trial is aimed to study the effect of oral use of lyophilized royal jelly for 4 weeks on immune system cytokine levels and cognitive functions in individuals aged 50-80 years without any neurological disease diagnosis.

Primary outcome measures are the Mini-Mental State Examination, the Alzheimer's Disease Assessment Scale-Cognitive Subscale, and the Geriatric Depression Scale.

Secondary outcome measures are serum interleukin-1β, interleukin-6, interleukin-10, tumor necrosis factor-α and transforming growth factor-β levels.

DETAILED DESCRIPTION:
Volunteers who apply to Bağcılar Medipol Mega University Hospital Neurology Polyclinic will be recruited, and their demographic information will be recorded.

Volunteers who meet eligibility criteria will be randomly divided into three groups considering age groups (50-64 years old and 65-80 years old).

Primary and secondary outcome measures will be evaluated in volunteers. The results obtained will be recorded.

Diet recommendations will be made to the volunteers for four weeks. The products detailed in the protocol will be used by the volunteers orally for four weeks on an empty stomach in the morning.

Primary and secondary outcome measures will be reassessed in volunteers on day 28. The results obtained will be recorded.

Obtained results will be evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 55 and 70,
* Male or female,

Exclusion Criteria:

* History of allergy to bee products
* Known history of lactose allergy
* Diagnosed dementia,
* MMSE score below 21,
* ADAS-Cog score of 12 and above,
* Body Mass Index of 35 and above,
* Be taking any medical medication, herbal product or dietary supplement for dementia, except for those who stopped using it at least 1 month before inclusion in our study,
* Being or having been treated for acute acquired brain injuries such as acute traumatic brain injury, acute onset stroke,
* Being followed up due to inflammatory disease,
* Diagnosis of chronic or acute infection,
* Taking corticosteroids or non-steroidal anti-inflammatory drugs,
* Being or having been treated for a psychotic illness,
* Severe anaemia, vital organ dysfunction or critical illness.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | Day 0
  The Turkish version of Mini-Mental State Examination, which has been tested for validity and reliability, will be administered by the same physician and at the same time interval.
Mini-Mental State Examination | Day 28
  The Turkish version of Mini-Mental State Examination, which has been tested for validity and reliability, will be administered by the same physician and at the same time interval.
Alzheimer's Disease Assessment Scale-Cognitive subscale | Day 0
  The Turkish version of Alzheimer's Disease Assessment Scale-Cognitive subscale, which has been tested for validity and reliability, will be administered by the same physician and at the same time interval.
Alzheimer's Disease Assessment Scale-Cognitive subscale | Day 28
  The Turkish version of Alzheimer's Disease Assessment Scale-Cognitive subscale, which has been tested for validity and reliability, will be administered by the same physician and at the same time interval.
Geriatric Depression Scale | Day 0
  The Turkish version of Geriatric Depression Scale, which has been tested for validity and reliability, will be administered by the same physician and at the same time interval.
Geriatric Depression Scale | Day 28
  The Turkish version of Geriatric Depression Scale, which has been tested for validity and reliability, will be administered by the same physician and at the same time interval.

SECONDARY OUTCOMES:
Serum Interleukin-1β Level | Day 0
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.
Serum Interleukin-1β Level | Day 28
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.
Serum Interleukin-6 Level | Day 0
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.
Serum Interleukin-6 Level | Day 28
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.
Serum Interleukin-10 Level | Day 0
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.
Serum Interleukin-10 Level | Day 28
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.
Serum Tumor Necrosis Factor-α Level | Day 0
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.
Serum Tumor Necrosis Factor-α Level | Day 28
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.
Serum Transforming Growth Factor-β Level | Day 0
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.
Serum Transforming Growth Factor-β Level | Day 28
  Measurement of serum levels will be done with the standard measurement method for the evaluation of inflammatory processes.